CLINICAL TRIAL: NCT02641210
Title: Impact of Periodontal Treatment on Serum Levels of Hepcidin and Hemoglobin: a Clinical Trial
Brief Title: Impact of Periodontal Treatment on Serum Levels of Hepcidin and Hemoglobin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Maranhao (Other)
Responsible Party: Principal Investigator, Sandra Augusta de Moura Leite, Professor in Federal University of Maranhao, Federal University of Maranhao
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23115-010215/2011-16
Record Dates: First submitted 2015-10-02; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis; Hepcidin; Hemoglobin; Inflammation
MeSH Terms: conditions — Chronic Periodontitis; Inflammation | interventions — Periodontal Index; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Periodontal Treatment (Experimental): The experimental group underwent nonsurgical periodontal therapy, performed by a single professional who performed the scaling and root planing procedures under local anesthesia using an ultrasonic device and Gracey and mini Gracey curettes, with Robson polishing brush and prophylactic paste. This therapy was performed in two sessions at seven day intervals, with no time limit, according to the needs of each periodontal condition. In each session, subjects received oral hygiene instruction (OHI) for use of toothbrushes for the modified Bass technique, dental floss and other complementary means (interdental brush, single tuft brush, electric toothbrush, etc.) when necessary. Supportive periodontal therapy was performed in 30, 60 and 90 days. Albendazole administration.
  Interventions: Procedure: Periodontal Treatment; Drug: Albendazole
- No Periodontal Treatment (No Intervention): Individuals in the control group underwent only the polishing of tooth surfaces with Robson brush and prophylactic paste fine-grained and topical fluoride application. After 90 days, they were reassessed with the same parameters of clinical examination of the baseline.

INTERVENTIONS:
Procedure: Periodontal Treatment — Periodontal Treatment using Gracey curettes and ultrasonic device.
  Other Names: Non-surgical Periodontal Therapy
  Arms: Periodontal Treatment
Drug: Albendazole — All participants took Albendazole 400 mg before the intervention.
  Other Names: drug administration
  Arms: Periodontal Treatment

SUMMARY:
Periodontitis is an inflammatory/infectious disease of high prevalence in the population and which has been linked to several chronic inflammatory systemic diseases. However, few studies have evaluated the periodontal disease in the absence of other inflammatory conditions stimulate inflammatory markers as C-reactive protein (CRP), Interleukin - 6 (IL-6) hepcidin and hemoglobin. The aim of this study was to evaluate the influence of nonsurgical periodontal therapy on the change of inflammatory markers and anemia in control subjects and patients with chronic periodontitis after three months.This interventional study included 67 individuals of both sexes, aged 30-65 years, without other diseases, except chronic periodontitis, with at least 20 teeth, selected from a total 125 individuals following the eligibility criteria. Periodontal clinical parameters (probing depth, bleeding on probing, clinical attachment level) and systemic, hematological as well as inflammatory markers CRP, IL-6 and hepcidin were compared before and after nonsurgical periodontal therapy by serum and plasma examination of control individuals and patients with chronic periodontitis.

DETAILED DESCRIPTION:
It conducted a non-randomized intervention study from April to October 2013, with individuals in the periodontics clinics of the Federal University of Maranhão State, São Luís, Brazil. The sample was selected from a total of 125 individuals, according to the eligibility criteria. Two groups were formed: experimental group (33 individuals) healthy patients except for the presence of chronic periodontitis in the advanced stage, and control group (30 subjects) patients without systemic disease proven by physical and biochemistry examination, and without chronic periodontitis.

The study was approved by the Ethics Committee on Human Research of the Federal University of Maranhão, São Luís, MA, Brazil under the protocol number 23115-010215 / 2011-16. All participants signed the consent form.

The sample size was defined on the basis of previous studies on the association between chronic periodontitis and systemic inflammatory markers.

All participants received an oral hygiene kit, attended a motivational speech with instructions on tooth brushing and flossing, and they were later referred for dental care.

At first visit, the medical record was checked for selecting volunteers without pre-diagnosed systemic diseases, in addition the general and periodontal clinical examination were performed, the urine collector was delivered, and drug intake [Albendazole 400 mg as a single dose]. After 15 days, subjects who met the initial selection criteria were sent for blood and urine collection for evaluation of biochemical markers. According to the results of laboratory tests, subjects were maintained or excluded after verification of those diagnosed with systemic diseases not previously identified.

The anamnesis and periodontal examination were carried out by a single trained examiner.It was collected the current and past medical and dental history, family history, social data, medications, possible changes of the menstrual flow, measurement of blood pressure, weight, height, and body mass index.

Oral clinical examination was also performed to diagnose the periodontal status of the participants. Then they were referred for dental care, according to their treatment needs.

After the therapy used, new clinical examination of the oral health of all participants was conducted 90 days after treatment. In the same period, new blood collection was performed for reassessment of biochemical markers.

The periodontal clinical examination used a periodontal probe type Williams in six sites per tooth (mesiobuccal, mid-buccal, it -vestibular, distolingual, medium-lingual, mesiolingual), performed by a single observer, dental surgeon, specialist in periodontics and previously trained. The intra-examiner concordance coefficient was 0.81 for probing depth and 0.77 for clinical attachment level. The following clinical parameters were evaluated: Probing depth (PD), gingival recession (GR), clinical attachment level (CAL), Visible Plaque Index (VPI), Bleeding on probing (BOP). This same examination at baseline was repeated 90 days after the initial examination and included the same clinical periodontal parameters.

Individuals who had at least two teeth with probing depth ≥ 5 mm and clinical attachment level ≥ 6 mm, associated with the presence of bleeding on probing, in the same site, 30 seconds after the first insertion probe, were diagnosed with periodontitis.

Blood samples (20ml) were collected in Ethylenediaminetetraacetic acid (EDTA) tubes after 12 hours fasting. The remainder of the EDTA-anticoagulated blood was centrifuged for 10 minutes at 3000 rpm to separate the plasma, aliquoted and stored at -70 until further analysis of the IL-6 concentrations.

The following laboratory tests were performed: total cholesterol, fasting glucose, triglycerides, albumin, glutamate oxalate transaminase, creatinine, uric acid, erythrocyte sedimentation rate (ESR), CRP, IL-6, Hepcidin, Serum Iron, Ferritin, Transferrin saturation, Blood parameters (hemoglobin, hematocrit, mean corpuscular volume - MCV, MCH), and urinalysis for abnormal elements and sediment (EAS).

Serum was obtained by addition of venous blood into a tube containing an activator of coagulation. After centrifugation for 15 minutes at 1800 rpm, the serum was separated. Serum was aliquoted piece for colorimetric evaluation of ferritin by chemiluminescence technique; serum iron and Ferrozine technique and transferrin saturation index, Goodwin's modified technique. The nephelometric was used for C-reactive protein of dosages and serum was stored at -70 °C remaining for analysis of hepcidin.

IL-6 and hepcidin were evaluated by the technique of immunoassay using ELISA kit, according to the manufacturer's instructions. Readings were made by automatic microplate reader and the absorbance was read at a wavelength of 450 nm in the spectrophotometer.

For statistical analysis, the investigators used a statistical software. Initially, there was a descriptive analysis through frequency measures, mean and standard deviation, median and interquartile range. Categorical variables were compared among groups using the chi-square test. The normal distribution of numerical variables was assessed Shapiro-Wilk test. The inferential analysis was made to assess the impact of the periodontal treatment on blood count variables, inflammatory markers, iron and periodontal parameters, used the paired Student's t test or the Wilcoxon test, and comparing the corresponding absolute delta between groups using the Mann-Whitney test. The significance level was set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Aged 30-65 years
* Without other chronic systemic diseases except periodontitis
* At least 20 teeth

Exclusion Criteria:

* Diabetes mellitus
* Congestive heart failure
* Chronic kidney disease
* Malignant neoplasms
* Acquired immunodeficiency syndrome
* Hypertension
* Pregnant women
* Nursing mothers
* Immunosuppressed by medication
* Women with changes in menstrual flow
* Smokers or ex-smokers for less than 10 years
* Usage history of NSAIDs or nonsteroidal and antibiotics within 3 months prior to the study and during the search
* Iron replacement in patients to treat anemia and carrying out subgingival scaling and periodontal surgery in 6 months prior to investigation.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in Hepcidin serum level after periodontal treatment as assessed by ELISA. | 90 days

SECONDARY OUTCOMES:
Changes in periodontal outcomes (Probing depth in millimeters and clinical attachment level in millimeter) after periodontal treatment. | 90 days
Percentage of sites with visible plaque and /or bleeding on probing after periodontal treatment. | 90 days
Changes in us-CRP serum level after periodontal treatment as assessed by ELISA. | 90 days
Changes in Interleukin 6 serum level after periodontal treatment as assessed by ELISA. | 90 days

OTHER OUTCOMES:
Changes in iron stores (Serum iron, ferritin and transferrin) after periodontal treatment. | 90 days